CLINICAL TRIAL: NCT02785861
Title: Evaluating the Effectiveness of Supervised Practice or Distance Supervised Physical Activity (Walking) in the Overall Management of Fatigue in Breast Cancer Patients During Hormonal Therapy: Pilot Study
Brief Title: Step by Step After Cancer
Acronym: SBSAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PI2012_843_0023
Record Dates: First submitted 2016-05-23; First posted 2016-05-30 (Estimated); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer
Keywords: hormonal therapy; walking; fatigue
MeSH Terms: conditions — Breast Neoplasms; Fatigue

ARMS (2):
- supervised practice (Experimental): brisk walking program twice a week over a period of 6 weeks, at an intensity of 60% of HR pic during 20 minutes.
  Biweekly session from 60% of the heart rate pic during 20 minutes will be proposed.
  Each patient of supervised walking group will meet the student each session
  Interventions: Behavioral: supervision of physical activity
- distance supervised physical activity (Experimental): brisk walking program twice a week over a period of 6 weeks, at an intensity of 60% of HR pic during 20 minutes.
  Biweekly session from 60% of the heart rate pic during 20 minutes will be proposed.
  Each patient of home-based walking group will be called by phone every week by the student to inform the patient of the progress of the training, collect the work and answer any questions
  Interventions: Behavioral: distance supervised physical activity

INTERVENTIONS:
Behavioral: supervision of physical activity
  Arms: supervised practice
Behavioral: distance supervised physical activity
  Arms: distance supervised physical activity

SUMMARY:
After treatment, women want to regain a 'normal' lifestyle while some factors interfere as chronic fatigue. In the absence of anemia, fatigue is often a consequence of physical deconditioning . The following protocol will focus at this problem.It will consist of a brisk walking program twice a week over a period of 6 weeks, at an intensity of 60% of HR pic during 20 minutes.

DETAILED DESCRIPTION:
Pinto and colleagues, for a walking level from 55 to 65% HRmax, estimated a reduction of fatigue in post treatment. Supervised exercise show greater adherence to short-term practice at home. However, there are a growing number of studies suggesting a practice at home, the most activity being walking. The authors do not justify the choice of the type of supervision. But physical activity with a professional and / or group in a specific place definitely has different effects in relation to practice at home. Segal and his colleagues in 2001 for the first time wished to compare the two types of supervision. The results are in favor of supervised exercise. The training was identical. However, to answer the five weekly sessions requested, the patient group had to complete two supervised practice sessions at home. So, the investigators really can not quantify the difference in impact between home practice and supervised practice. In a meta-analysis, Velthuis and colleagues conclude a significant difference in fatigue during treatment for a supervised aerobic exercise against a home that does not show significant difference. If the training is the same in both situations, the investigators should not find any difference in physiologic responses. However, the psychological impact can vary from one situation to another.

The following protocol will focus at this problem. It will consist of a brisk walking program twice a week over a period of 6 weeks, at an intensity of 60% of HR pic during 20 minutes.

Biweekly session from 60% of the heart rate pic during 20 minutes will be proposed.

Each patient of supervised walking group will meet the student each session. Each patient of home-based walking group will be called by phone every week by the student to inform the patient of the progress of the training, collect the work and answer any questions.

ELIGIBILITY:
Inclusion Criteria:

* Sex: female
* Age less than or equal to 75 years
* Breast cancer stage I to III
* Chemotherapy and / or radiotherapy adjuvant completed
* Hormone treatments ongoing

Exclusion Criteria:

* Age over 75 years
* Breast cancer stage IV and O
* Anemia, Cardiac arrhythmia, asthma, hypertension or uncontrolled diabetes, coronary artery disease or severe respiratory disease, psycho-cognitive may disturb walking program

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2013-02-18 (Actual); Primary Completion 2026-02-10 (Actual); Study Completion 2026-02-10 (Actual)

PRIMARY OUTCOMES:
fatigue of the patient with QLQC-30 | 6 weeks

SECONDARY OUTCOMES:
Global Quality of life with QLQC-30 | 6 weeks
Activity level with IPAQ | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu BOONE, MD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France